CLINICAL TRIAL: NCT04218552
Title: A Randomized, Double-Blind, Parallel, Multi-Center, Phase 2 Clinical Trial to Determine the Optimal Dose of AD-209 in Patients With Essential Hypertension
Brief Title: Determining the Optimal Dose of AD-209 in Patients With Essential Hypertension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Addpharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AD-209P2
Record Dates: First submitted 2020-01-03; First posted 2020-01-06 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-01

CONDITIONS: Hypertension,Essential
MeSH Terms: conditions — Essential Hypertension | interventions — Telmisartan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Experimental 1 (Experimental): AD-209 High
  Interventions: Drug: AD209
- Experimental 2 (Experimental): AD-209 Middle
  Interventions: Drug: AD209
- Experimental 3 (Experimental): AD-209 Low
  Interventions: Drug: AD209
- Active Comparator 1 (Active Comparator): Amlodipine Low
  Interventions: Drug: Amlodipine low
- Active Comparator 2 (Active Comparator): Amlodipine High
  Interventions: Drug: Amlodipine high
- Active Comparator 3 (Active Comparator): Telmisartan
  Interventions: Drug: Telmisartan
- Placebo comparator (Placebo Comparator): Placebo
  Interventions: Drug: AD209; Drug: Amlodipine low; Drug: Amlodipine high; Drug: Telmisartan

INTERVENTIONS:
Drug: AD209 — PO, Once daily(QD), 8weeks
  Other Names: AD209 Placebo
  Arms: Experimental 1; Experimental 2; Experimental 3; Placebo comparator
Drug: Amlodipine low — PO, Once daily(QD), 8weeks
  Other Names: Amlodipine low placebo
  Arms: Active Comparator 1; Placebo comparator
Drug: Amlodipine high — PO, Once daily(QD), 8weeks
  Other Names: Amlodipine high placebo
  Arms: Active Comparator 2; Placebo comparator
Drug: Telmisartan — PO, Once daily(QD), 8weeks
  Other Names: Telmisartan placebo
  Arms: Active Comparator 3; Placebo comparator

SUMMARY:
The purpose of this study is to determine the optimal dose of AD-209 in patients with Essential Hypertension.

DETAILED DESCRIPTION:
Condition or disease : hypertension Intervention/treatment Drug : AD-209-H Drug : AD-209-M Drug : AD-209-L Drug : Placebo Drug : Amlodipine Drug : Telmisartan Phase : Phase 2

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Other inclusions applied

Exclusion Criteria:

* orthostatic hypotension with symptom
* Other exclusions applied

Ages: 19 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2020-02-25 (Actual); Primary Completion 2021-02-25 (Actual); Study Completion 2021-02-25 (Actual)

PRIMARY OUTCOMES:
1. Change rate of MSSBP | [ Time Frame: baseline, 8 weeks ]
  Change from baseline in mean sitting systolic blood pressure

SECONDARY OUTCOMES:
1. Change rate of MSSBP | [ Time Frame: baseline, 4 weeks ]
  Change from baseline in mean sitting systolic blood pressure
2. Change rate of MSDBP | [ Time Frame: baseline, 4 weeks, 8 weeks ]
  Change from baseline in mean sitting diastolic blood pressure
3. Proportion of BP normalization MSSBP/MSDBP < 140/90 mmHg MSSBP/MSDBP < 130/80 mmHg (Diabetes or Chronic renal disease) | [ Time Frame: 4 weeks, 8 weeks ]
  Proportion of subjects achieving blood pressure control
4.Reaction rate of BP | [ Time Frame: baseline, 4 weeks, 8 weeks ]
  Proportion of reduction from baseline in MSSBP/MSDBP ≥ 20/10 mmHg

CONTACTS AND LOCATIONS:
Overall Officials: ChangGu Park, M.D., Ph.D, Principal Investigator — Korea University Guro Hospital
Locations (1):
- Korea University Guro Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sung KC, Sung JH, Cho EJ, Ahn JC, Han SH, Kim W, Kim KH, Sohn IS, Shin J, Kim SY, Kim KI, Kang SM, Park SJ, Kim YJ, Shin JH, Park SM, Park CG. Efficacy and safety of low-dose antihypertensive combination of amlodipine, telmisartan, and chlorthalidone: A randomized, double-blind, parallel, phase II trial. J Clin Hypertens (Greenwich). 2022 Oct;24(10):1298-1309. doi: 10.1111/jch.14570. Epub 2022 Sep 12. PMID 36094783